CLINICAL TRIAL: NCT01968252
Title: Validation of Speckle-tracking Echocardiography Measurements of Tricuspid Annular Plane Systolic Excursion During Transesophageal Echocardiography
Brief Title: Speckle-tracking Tricuspid Annular Plane Systolic Excursion
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0107-14-EP
Record Dates: First submitted 2013-10-16; First posted 2013-10-23 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Function, Right
Keywords: Speckle-tracking echocardiography; Transthoracic echocardiography; Transesophageal echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intraoperative Patient: All patients in the cohort will be scheduled to undergo a planned surgical procedure in which the subject will undergo general anesthesia and the procedure and/or the patient will require transesophageal echocardiographic monitoring for the procedure.
  Interventions: Other: Concurrent TTE and TEE

INTERVENTIONS:
Other: Concurrent TTE and TEE — All subjects will undergo both transthoracic echocardiography and transesophageal echocardiography to compare the results of measurements obtained from both imaging locations.

SUMMARY:
The study is designed to validate the use of speckle-tracking echocardiography to measure tricuspid annular plane systolic excursion as a measurement of right ventricular function during transesophageal echocardiography.

DETAILED DESCRIPTION:
1. Use of speckle-tracking echocardiography to validate tricuspid annular plane systolic excursion measurements with transesophageal echocardiography.
2. This study intends to validate the use of speckle-tracking echocardiography to measure the distance the tricuspid annulus moves during the systolic phase. The guideline articles regarding right ventricular function suggest m-mode measurements from the transthoracic approach and the same measurements may underestimate the actual distance on transesophageal echocardiography. This speckle-tracking technology will allow this distance to be measured despite its often non-parallel motion to the ultrasound beam, which otherwise limits the reliability of the valve recorded.
3. All subjects undergoing a planned surgical procedure in which the use of transesophageal echocardiography would be used regardless for their management.
4. No interventions, only evaluation of the measurements obtained with transthoracic echocardiography compared to transesophageal echocardiography.
5. No follow-up, study will be completed at the time of image acquisition.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who are scheduled to undergo general anesthesia and concurrently will be managed with intraoperative transesophageal echocardiography will be included in potential subjects.

Exclusion Criteria:

* Subjects who do not have adequate transesophageal and/or transthoracic imaging windows to allow for accurate analysis of tricuspid annular motion.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be scheduled to undergo a surgical procedure requiring general anesthesia and either due to subject factors or procedure factors, the use of intraoperative transesophageal echocardiographic monitoring will occur. These subjects will then have both transesophageal and transthoracic echocardiographic measurements of one variable of right ventricular function to validate the results from the transesophageal window.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Speckle-tracking derived tricuspid annular plane systolic excursion with transesophageal echocardiography | 1 hour
  Speckle-tracking derived tricuspid annular plane systolic excursion with transesophageal echocardiography

SECONDARY OUTCOMES:
M-mode derived tricuspid annular plane systolic excursion with transesophageal echocardiography | 1 hour
  M-mode derived tricuspid annular plane systolic excursion with transesophageal echocardiography
M-mode derived tricuspid annular plane systolic excursion with transthoracic echocardiography | 1 hour
  M-mode derived tricuspid annular plane systolic excursion with transthoracic echocardiography
Speckle-tracking derived tricuspid annular plane systolic excursion with transthoracic echocardiography | 1 hour
  Speckle-tracking derived tricuspid annular plane systolic excursion with transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas W Markin, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Ahmad H, Mor-Avi V, Lang RM, Nesser HJ, Weinert L, Tsang W, Steringer-Mascherbauer R, Niel J, Salgo IS, Sugeng L. Assessment of right ventricular function using echocardiographic speckle tracking of the tricuspid annular motion: comparison with cardiac magnetic resonance. Echocardiography. 2012;29(1):19-24. doi: 10.1111/j.1540-8175.2011.01519.x. Epub 2011 Oct 4. PMID 21967480
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Mor-Avi V, Lang RM, Badano LP, Belohlavek M, Cardim NM, Derumeaux G, Galderisi M, Marwick T, Nagueh SF, Sengupta PP, Sicari R, Smiseth OA, Smulevitz B, Takeuchi M, Thomas JD, Vannan M, Voigt JU, Zamorano JL. Current and evolving echocardiographic techniques for the quantitative evaluation of cardiac mechanics: ASE/EAE consensus statement on methodology and indications endorsed by the Japanese Society of Echocardiography. J Am Soc Echocardiogr. 2011 Mar;24(3):277-313. doi: 10.1016/j.echo.2011.01.015. PMID 21338865